CLINICAL TRIAL: NCT05799703
Title: Effect Of Reciprocal Electrical Stimulation Versus Kinesio Taping On Hand Functions In Hemiparetic Cerebral Palsy Children
Brief Title: Reciprocal Electrical Stimulation Versus Kinesio Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basma Elsaid Mahmoud Bakr (Other)
Responsible Party: Sponsor-Investigator, Basma Elsaid Mahmoud Bakr, Effect Of Reciprocal Electrical Stimulation Versus Kinesio Taping On Hand Functions In Hemiparetic Cerebral Palsy Children, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EG, KFS lab Research 6
Record Dates: First submitted 2023-03-03; First posted 2023-04-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: kinesio taping; reciprocal electrical stimulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): will receive RES in addition to the traditional exercise program.
  Interventions: Device: electrical stimulation device
- Group (B) (Active Comparator): will receive KT in addition to the traditional exercise program.
  Interventions: Other: kinesio taping

INTERVENTIONS:
Device: electrical stimulation device — the device has 2 channels ,4 electrodes with multiple ems programs
  Arms: Group (A)
Other: kinesio taping — kinesio tape a therapeutic tape that's applied strategically to the body to provide support, lessen pain, reduce swelling, and improve performance
  Arms: Group (B)

SUMMARY:
This study will be conducted to:

1. evaluate the effect of kinesio taping on hand functions in hemiplegic cerebral palsy children
2. compare between the effects of reciprocal electrical stimulation and kinesio taping on hand functions in hemiplegic cerebral palsy children.

DETAILED DESCRIPTION:
A. Patients preparation All the children demographic and outcome measures data will be collected in specially well-designed sheets1. Evaluation of fine motor skills using PDMS-2 Evaluation of hand function using Besta scale

. The traditional exercise program (given to both groups):

1. Treatment protocol in Group A, Reciprocal electrical stimulation protocol

   * The device has two channels that can stimulate two opposing groups of muscles alternatively (reciprocate).
   * During ES, the child sits in a chair with his treated forearm resting on a pillow placed on the bed in front of him.
   * The electrodes will be placed as follows:
   * Channel 1 (stimulates wrist and hand extensors) electrodes placed over the dorsum of the forearm as follows: the active electrode is placed over the common extensor origin, while in different over the motor point of extensor pollicis longus, abductor pollicis longus, and extensor indices.
   * Channel 2 (stimulates wrist and hand flexors) electrodes placed on the palmar side of the forearm are as follows: the negative electrode is placed between the finger flexors and wrist flexors. The positive electrode is placed over the tendonportion of the forearm,
   * The treatment duration will be 20 minutes.
   * The treatment protocol will be repeated 3 times per week for 12 weeks.
2. Treatment protocol in Group B, Kinesio taping protocol:

   * Kinesio taping will be applied on both sides of the upper limb.
   * The applied area will be from the proximal one-third of the forearm to the wrist and then will be split into 5 straps into the distal interphalangeal joint of fingers.
   * On the dorsal side, KT will be applied on the forearm, wrist, and fingers extensors for improvement of wrist and fingers extension.
   * On the plantar side, KT will be applied on the forearm, wrist, and fingers flexors for inhibition of wrist and fingers flexion.
   * Taping will be applied for 6 days, 24 h a day, on the affected upper limb, and it will be removed for only one day per week.

ELIGIBILITY:
Inclusion Criteria:

* A medical diagnosis of spastic hemiplegic CP made by paediatricians or pediatric neurologists.
* Children with spasticity grades ranged from 1 to 1+ according to MAS.
* Their age range from 4 to 6 years.
* Children who can sit on the chair with good balance and recognize and follow verbal orders and commands included in both testing and training techniques

Exclusion Criteria:

* They had a permanent deformity (bony or soft tissue contractures).
* Children having visual or auditory defects.
* Children with intelligence quotient less than 70.
* Children who had Botox application to the upper extremity in the past 6 months or had undergone a previous surgical intervention to wrist and hand.
* A history of epileptic seizure and any diagnosed cardiac or orthopaedic disability that may prevent the use of assessment methods.
* Children who are absent in two taping change sessions

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Fine motor skills | 3 months
  we will use Peabody developmental motor scale-2 to assess fine motor skills

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafrelsheikh, Egypt